CLINICAL TRIAL: NCT06344572
Title: A Multicenter, Randomized, Open-label, Controlled Pivotal Study to Evaluate the Efficacy and Safety of Software SAT-001 in Slowing Myopia Progression and Treatment in Pediatric Patients With Myopia
Brief Title: Pivotal Study of SAT-001 in Treatment of Pediatric Patient With Myopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAT001-KP-002
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAT-001 (Experimental): SAT-001(Software as Medical Device)+single vision spectacles
  Interventions: Device: SAT-001
- Single vision spectacles (Active Comparator): Wearing single vision spectacles
  Interventions: Other: Single vision spectacles

INTERVENTIONS:
Device: SAT-001 — Device: SAT-001(a Software as Medical Device) Using SAT-001 application for 48 weeks and wearing single vision spectacles
  Arms: SAT-001
Other: Single vision spectacles — Wearing single vision spectacles
  Arms: Single vision spectacles

SUMMARY:
The objective of this clinical investigation is to evaluate the efficacy and safety of SAT-001 designed as Software as Medical Device (SaMD) for slowing myopia progression and treatment in pediatric myopia patients.

DETAILED DESCRIPTION:
Myopia is a common refractive error affecting approximately 30 % of the global population, with even higher prevalence in Asian countries including Korea. This study is a confirmatory clinical trial designed to evaluate the efficacy and safety of SAT-001 for slowing the progression of myopia in children, based on the results of the exploratory clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5 to less than 9
2. Meet the following refractive criteria by cycloplegic refraction

   1. Spherical equivalent refractive error (SER): -0.75 to less than -6.00 D in each eye
   2. Astigmatism of 1.50 D or less in each eye
   3. Anisometropia of 2.00 D or less
3. Best corrected visual acuity of 0.2 logMAR or better in each eye at the Screening Visit
4. Able to successfully accomplish SAT-001, the investigational device (able to follow the written and verbal instruction)
5. Subjects and their legal guardians who agree to participate in the clinical trial and are willing to provide the signed informed consent after receiving and comprehending the explanation of the description of this clinical trial (subject under 6 can make a mark for agreement after full information and understanding)

Exclusion Criteria:

1. History of atropine use within 3 days prior to Baseline (Visit 2) (prior treatment of myopia control with low dose atropine within 1 month prior to Baseline)
2. Current or prior use of multifocal lenses (e.g. progressive addition lenses), orthokeratology (Ortho-K, e.g. Dream lens), or Rigid gas permeable (RGP) within 1month prior to Baseline(Visit 2)
3. Ocular abnormalities in cornea, lens, central retina, iris, ciliary body, etc., or presence of malignant tumors in the orbital area
4. History of eye diseases such as manifest strabismus, intermittent strabismus, amblyopia, and nystagmus (excluding strabismus that maintains binocular vision)
5. History of ocular surgery such as eyelid surgery, strabismus surgery, intraocular surgery, or refractive correction surgery (excluding simple double eyelid surgery)
6. Down's syndrome or cerebral palsy
7. Within 6 months prior to the Screening visit (Visit 1), has experience of other clinical trial medications or investigational device
8. Clinically significant systemic diseases such as congenital heart disease, respiratory disease, endocrine disease, and neurological disease that the investigator may consider inappropriate for participation in the clinical trials
9. Systemic diseases that could impact both vision and visual field
10. History of growth hormone treatment within 1 month prior to Baseline (Visit 2)
11. Other reasons for participation in the trial at the discretion of the investigator

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Axial Length | Baseline, 48weeks

SECONDARY OUTCOMES:
Change in Axial Length | Baseline, 12weeks, 24weeks, 36weeks
Change in cycloplegic Spherical Equivalent Refractive Error | Baseline, 24weeks, 48weeks
Change in cycloplegic Spherical Equivalent Refractive Error relative to baseline depending on the myopia severity(mild myopia, moderate myopia) | Baseline, 24 weeks, 48 weeks
Change in axial length relative to baseline depending on the myopia severity(mild myopia, moderate myopia) | Baseline, 12weeks, 24weeks, 36weeks, 48weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Paik HJ, Lee BJ, Lim DH, Han SY, Jung EH, Shin HJ, Kim HK, Kim US, Kim WJ, Choi HY, Park J, Rhiu S, Lee J, Kim M, Kim K. Digital therapeutics approach for young children with myopia using SAT-001 (DAYS): study protocol for a randomized controlled trial. Trials. 2025 Apr 8;26(1):128. doi: 10.1186/s13063-025-08717-w. PMID 40200346